CLINICAL TRIAL: NCT01302236
Title: Effects of Eplerenone on Blood Pressure, Heart and Kidney in Elderly Hypertensive Early Stage Chronic Kidney Disease Patients
Brief Title: Effect of Eplerenone in Elderly Hypertensive Early Stage Chronic Kidney Disease (CKD) Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We could not find patients who agreed to enrolled this clinical study.
Sponsor: Jichi Medical University (Other)
Responsible Party: Principal Investigator, Yoshiyuki Morishita, MD. PhD, Jichi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMU-N2
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension; Chronic Kidney Disease.
Keywords: Elderly; Early stage chronic kidney disease; Hypertension; Eplerenone
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eplerenone (Experimental)
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — 50mg/day for all as initial dose, 100mg/day for the patients that still show hypertension(above 140/90mmHg)after one month 150mg treatment,oral,on 6 months
  Other Names: Selective aldosterone blocker

SUMMARY:
The purpose of this study is to determine whether eplerenone is effective in the treatment of blood pressure, heart function, renal function in elderly hypertensive stage1 (eGFR>=90ml/min/1.73m2) and stage2 (eGFR 60-89ml/min/1.73m2) chronic kidney disease (CKD) patients.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) was reported to be affecting 11% of the all population. This number is much higher in the elderly population and may be as high as 30%. CKD is an independent risk factor of cardiovascular disease (CVD). This is called "Cardio-renal Continuum". The renin-angiotensin-aldosterone system (RAS) plays pivotal roles in both cardiovascular and renal functions.

The increased oxidative stress by activated RAS on vascular endothelium is one of important factor to development of Cardio-renal Continuum. The blockade of RAS by angiotensin I converting enzyme inhibitors (ACEIs) and/or angiotensin receptor blockers (ARBs) has been reported to ameliorate the renal disease and CVD; however,they do not completely suppress RAS and may induce aldosterone breakthrough that plays important roles for the development of CVD. Eplerenone, a selective aldosterone blocker, is effective against essential hypertension; however, little is known about the effects of eplerenone on heart and kidney functions in elderly hypertensive CKD patients. In this study, we assessed the efficacy of eplerenone on heart and kidney functions in elderly hypertensive early stage (stage1 (eGFR>=90ml/min/1.73m2) and stage2 (eGFR 60-89ml/min/1.73m2)) CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stage1(eGFR>=90ml/min/1.73m2) and stage2 (eGFR 60- 89ml/min/1.73m2)chronic kidney disease
* Clinical diagnosis of Hypertension (Blood pressure >=140/90mmHg)
* Elderly people(>=65 years old)

Exclusion Criteria:

* The patients who are already taking eplerenone
* Stage3(eGFR 30-60 ml/min/1.73m2),stage4(eGFR 15-30 ml/min/1.73m2)and stage5 (eGFR <15 ml/min/1.73m2) CKD patients
* The patients who are receiving hemodialysis or peritoneal dialysis
* The patients who are taking itraconazole, ritonavir and nelfinavir
* The patients who are taking potassium-sparing diuretics and potassium supplement
* The patients who have hyperkalemia(>=5.5mEq/ml)
* Severe heart failure (>=NYHA class III)
* Insulin dependent diabetic mellitus or poor controlled insulin independent diabetic mellitus (>=HbA1c 9.0&)
* Severe liver dysfunction (five folds increased AST or ALT than standard values)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The change of heart function confirmed by echocardiograph and plasma level of BNP | 6 months
The change of renal function confirmed by eGFR and proteinuria. | 6 months

SECONDARY OUTCOMES:
The change of blood pressure | 6 months
  The change of systolic blood pressure and diastolic blood pressure
The change of oxidative stress markers confirmed by plasma level of 8-OHdG and d-ROM | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiyuki Morishita, MD. PhD, Principal Investigator — Division of Nephrology, Department of Medicine, Jichi Medical University

REFERENCES:
- [Background] Morishita Y, Hanawa S, Chinda J, Iimura O, Tsunematsu S, Kusano E. Effects of aliskiren on blood pressure and the predictive biomarkers for cardiovascular disease in hemodialysis-dependent chronic kidney disease patients with hypertension. Hypertens Res. 2011 Mar;34(3):308-13. doi: 10.1038/hr.2010.238. Epub 2010 Dec 2. PMID 21124333